CLINICAL TRIAL: NCT03863873
Title: Platelet-Rich Plasma in the Treatment of Patients With Idiopathic Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Reham Magdy, Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRPCTS
Record Dates: First submitted 2019-02-16; First posted 2019-03-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Platelet-rich plasma
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP Injection Group (Active Comparator): PRP Preparation: 16 ml of blood was obtained from each patient using special PRP kits (GD medical pharma, Dutch company). The blood was collected on citrated tubes with a mixing ratio of 9:1 by volume. Tubes underwent 1st centrifugation at speed of 3000 rpm (704g) for 3 minutes (to separate red blood cells from plasma). Plasma was then removed by syringe and then placed into another sterile tube with no anticoagulant and then underwent 2nd centrifugation at speed of at 4000 rpm (1252g) for 15 min. The supernatant platelet-poor plasma was then removed leaving 2 ml of PRP pellets in the sediment, and suspend the PRP pellets by gentle shaking of the tube. PRP is activated by adding 200 μl of 0.025 calcium chloride(Dhurat and Sukesh, 2014).
  Interventions: Procedure: Platelet-Rich Plasma Injection Group
- Steroid injection Group (Active Comparator): A single injection of methylprednisolone acetate 40 mg/ml using a technique similar to that described for the PRP injection
  Interventions: Procedure: Platelet-Rich Plasma Injection Group

INTERVENTIONS:
Procedure: Platelet-Rich Plasma Injection Group — Platelet-Rich Plasma Injection Group

SUMMARY:
This is a randomized controlled trial in a cohort of Egyptian patients suffered from mild to moderate idiopathic carpal tunnel. They were randomly divided into two groups. Group 1: patients received ultrasound-guided platelet-rich plasma injection and group 2 patients received ultrasound-guided corticosteroid injection. The outcome measures were assessed via Visual Analogue Scale, the Boston Carpal Tunnel Syndrome Questionnaire, electrophysiological findings in sensory and motor function of the median nerve and morphological changes of median nerve detected by ultrasound.

DETAILED DESCRIPTION:
Intervention:

PRP Injection Group(PRP-inj-G) - This group included 49 patients (40 females and 9 males). Their age ranged from 20 to 60 years.

PRP Preparation: 16 ml of blood was obtained from each patient using special PRP kits (GD medical pharma, Dutch company). The blood was collected on citrated tubes with a mixing ratio of 9:1 by volume. Tubes underwent 1st centrifugation at speed of 3000 rpm (704g) for 3 minutes (to separate red blood cells from plasma). Plasma was then removed by syringe and then placed into another sterile tube with no anticoagulant and then underwent 2nd centrifugation at speed of at 4000 rpm (1252g) for 15 min. The supernatant platelet-poor plasma was then removed leaving 2 ml of PRP pellets in the sediment, and suspend the PRP pellets by gentle shaking of the tube. PRP is activated by adding 200 μl of 0.025 calcium chloride(Dhurat and Sukesh, 2014).

Ultrasound-Guided Injection: Proper preparation with an antiseptic solution of skin overlying the point of injection was performed guided by ultrasonography (Siemens Acuson P300 machine). With the palm facing upward and the wrist joint in slight extension, the MN will be recognized at the inlet of the CT(Wu et al., 2017). The injection was guided by ultrasound with the use of the ulnar in-plane technique(Lee et al., 2014). Ulnar artery was identified by the means of Doppler imaging, and a 25-gauge needle was introduced from the ulnar side of the wrist between CT and MN. Then the entire CT was scanned to confirm that the injection had dispersed through the proximal to the distal area of the CT. All patients were observed for 30 minutes post-injection for the possibility of dysesthesia or bleeding(Wu et al., 2017).

PRP injection: A 25-gauge needle was gently introduced one cm proximal to the distal wrist-flexion crease just to the ulnar side of the palmaris longus tendon and 2 ml of PRP was injected into the CT.

Steroid injection Group(St-inj-G) - included 49 patients (41 females and 8 males)with their age ranged from 20 to 60 years. A single injection of methylprednisolone acetate 40 mg/ml using a technique similar to that described for the PRP injection

Post-injection care for both groups:

* Some patients may have minimal to moderate discomfort after injection. So, to control pain, patients should apply ice on the injection site and also modify activity as tolerated.
* Rest for one day.
* The patient immediately returns to work two days after injection.
* Pain medication in the form of paracetamol only was allowed for the next 3 months if needed. The patients were instructed to stop analgesics 48 hours before the visit to allow proper symptoms assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild-to-moderate idiopathic CTS with clinical manifestations failed to respond to conservative treatment ( such as splint, medications, Physical therapy) for at least 3 months and they were diagnosed by electrophysiological study and musculoskeletal ultrasound.

Exclusion Criteria:

* Diabetes
* Hypothyroidism
* Rheumatoid arthritis
* Previous carpal tunnel decompressive surgery
* Cervical radiculopathy, polyneuropathy, brachial plexopathy, traumatic nerve injury, thoracic outlet syndrome
* Previous corticosteroid injection into the carpal tunnel in the preceding 4 weeks
* Anemia (hemoglobin <10gm%)
* Coagulopathy
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Pain improvement | three months
  The VAS-pain score is composed of a continuous horizontal line. This line is 100 mm in length. To measure the intensity of pain, the score is anchored by (0 score = no pain) at one end and (100 score = worst imaginable pain) on the other end. The patient places a mark to the VAS line at the point which represents the intensity of his pain.
Function improvement | three months
  The Boston CT Questionnaire (BCTQ) is a patient-based outcome measure that was designed specifically for CTS patients. BCTQ has 2 distinct scales, the Symptom Severity Scale (BCTQ-SSS) containing 11 questions and the Functional Status Scale (BCTQ-FSS) containing 8 items. All questions were rated for degree of difficulty on a 5points scale. Each scale producesa final average score (sum of the scores divided by number of items) with a higher score indicative of greater disability. The BCTQ was used as an outcome measure in clinical trials, and has been reported as a validity and reliable tool for assessment of CTS.
Edema | three months
  US examination of the m-CSA for all patients was performed using a 7-13 MHz linear array probe with a calibrated device (Siemens, Acuson P300 apparatus) on the same day of EDX examination and clinical evaluation. All US examinations were performed with the wrists at the neutral position. The US examiner applied a minimal pressure force to avoid induction of artificial nerve deformation. Three measurements of the m-CSA at the level of most-protuberant portion of the pisiform bone were performed. The mean of the three measurements is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Senna MK, Shaat RM, Ali AAA. Platelet-rich plasma in treatment of patients with idiopathic carpal tunnel syndrome. Clin Rheumatol. 2019 Dec;38(12):3643-3654. doi: 10.1007/s10067-019-04719-7. Epub 2019 Aug 16. PMID 31420812